CLINICAL TRIAL: NCT00017199
Title: Phase II Study of PS-341 in Metastatic Neuroendocrine Tumors
Brief Title: PS-341 in Treating Patients With Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068660; OSU-00H0328; NCI-1856
Record Dates: First submitted 2001-06-06; First posted 2004-02-16 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2007-05

CONDITIONS: Gastrointestinal Carcinoid Tumor; Islet Cell Tumor
Keywords: metastatic gastrointestinal carcinoid tumor; gastrinoma; insulinoma; somatostatinoma; glucagonoma
MeSH Terms: conditions — Adenoma, Islet Cell; Gastrinoma; Insulinoma; Somatostatinoma; Glucagonoma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of PS-341 in treating patients who have metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate of patients with metastatic neuroendocrine tumors treated with bortezomib.
* Determine the toxicity of this drug in this patient population.
* Determine the pharmacodynamics to correlate proteasome inhibition and efficacy of this drug in this patient population.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for at least 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond CR.

PROJECTED ACCRUAL: A total of 16-25 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic carcinoid tumor or islet cell tumor

  * Well-differentiated neuroendocrine tumor OR
  * Well-differentiated neuroendocrine carcinoma
* Measurable disease in at least 1 dimension

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are considered nonmeasurable:

    * Lesions in a previously irradiated area
    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed
    * Cystic lesions

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* Leukocyte count at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other uncontrolled illness
* No ongoing active infection
* No psychiatric illness or social situation that would preclude study
* No history of allergic reaction to compounds of similar chemical or biologic composition to bortezomib
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy (interferon alfa)

Chemotherapy:

* No more than 1 prior systemic chemotherapy regimen (except hepatic artery chemoembolization)
* At least 4 weeks since prior systemic chemotherapy (6 weeks for nitrosoureas)
* At least 12 weeks since prior hepatic artery chemoembolization (unless liver lesions are not indicator lesions)
* Stable dose long-acting octreotide therapy (Sandostatin LAR) within the past 3 months allowed
* Concurrent subcutaneous octreotide for breakthrough symptomatic relief allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agents, commercial agents, or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha H. Shah, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio